CLINICAL TRIAL: NCT05063877
Title: A Dose-Ranging Safety, Tolerability, and Exploratory Efficacy Study of Adjunctive EQU-001 for Seizures in Adults With Epilepsy
Brief Title: Safety, Tolerability, and Exploratory Efficacy of Adjunctive EQU-001 for Seizures in Adults With Epilepsy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Equilibre Biopharmaceuticals B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EQU-201
Record Dates: First submitted 2021-09-22; First posted 2021-10-01 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Epilepsy
Keywords: Epilepsy; Seizure; Adult
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Intervention Model Description: 4:1 treatment to placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All parties are blinded for the initial two week safety period. A sponsor study physician and statistician (not an outcomes assessor) will be unblinded after the initial two week period to monitor ongoing safety, PK and concomitant drug levels
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Matched placebo control 10 mg capsule or 20 mg capsules totaling to 10 mg, 20 mg, 40mg or 60 mg will be administered once daily orally for 12 weeks with the option for open-label extension.
  Intervention: Drug: Placebo
  Interventions: Drug: Placebo
- Study drug EQU-001 (Experimental): 10mg capsules or 20 mg EQU-001 capsules totally 10 mg, 20 mg, 40 mg, 60 mg will be administered once orally daily to active-treatment subjects for 12-weeks with the option for open-label extension. During the open-label extension, subjects taking 60 mg dose for 4 weeks or longer may increase to 80 mg per day dose, at the discretion of the PI.
  Intervention: Drug : EQU-001
  Interventions: Drug: EQU-001

INTERVENTIONS:
Drug: Placebo — Matched placebo
  Arms: Placebo
Drug: EQU-001 — EQU-001 in 10 mg and 20 mg capsules
  Arms: Study drug EQU-001

SUMMARY:
This is a double-blind, placebo controlled, randomized study of dose-ranging safety, tolerability, exploratory efficacy of adjunctive EQU-001 for seizures using the continuous reassessment method in patients diagnosed with epilepsy.

DETAILED DESCRIPTION:
EQU-201 is a Phase 2 randomized, double-blind, placebo-controlled study to evaluate dose-ranging safety, tolerability, and exploratory efficacy of adjunctive EQU-001 using the continuous reassessment method (CRM). 10 participants diagnosed with epilepsy according to the International League Against Epilepsy (ILAE) Classification of the Epilepsies 2017 criteria whose seizures are uncontrolled on one to four concomitant antiepileptic drugs (AEDs) for ≥4 weeks will be enrolled in 4 dose cohorts (10 mg, 20 mg, 40 mg, 60 mg) The participants will be randomized 4:1, drug to placebo. The dosing is for 12 weeks, after which, safety data will be reviewed post 14 days to determine whether the next cohort can be opened. Once the 12-week study dosing period is complete, all subjects may enroll in an open-label extension, during which period investigators may make dose adjustments down to 20 mg and up 80 mg.

This study of EQU-001 will provide safety of a range of doses, tolerability, and PK data in patients with epilepsy and aims to identify drug-specific DLTs and MTD. The PK component will characterize the PK of EQU-001 to inform dosing and may help to correlate exposures with any DLTs or other treatment-related AEs. The open label extension component will provide data on subject safety, tolerability and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide informed consent, or consent provided by a Legally Authorized Representative (LAR)
2. Diagnosed with epilepsy according to ILAE 2017 criteria and with uncontrolled countable seizures (as per Epilepsy Study Consortium review) on one to four concomitant anti-seizure medicines (AEDs) at optimal stable dosages for at least 4 weeks prior to screening and throughout the treatment period
3. Age 18 to 60 years of age
4. Must have had a brain MRI or CT scan with an available report (images need not be available) that is negative for other confounding conditions
5. Must have an EEG report consistent with the subject's seizure type(s)
6. Pre-menopausal females and males with pre-menopausal sexual partners should either be sexually inactive (abstinent) for 21 days prior to the first dose, throughout the study, and for 14 days following the last dose or, if heterosexually active, agree to use of one of the following acceptable birth control methods for the period above:

   1. Intrauterine device (IUD) in place
   2. Hormonal contraceptives plus barrier method
   3. At least 2 barrier methods (condom, diaphragm) with spermicide
   4. Surgical sterilization of participant or partner(s) (bilateral tubal ligation, hysterectomy, bilateral oophorectomy, vasectomy > 6 months ago)
7. Able and willing to adhere to protocol; the subject or selected observer can keep an accurate seizure diary
8. Before progressing from Baseline Period to Randomization:

   1. A subject must experience at least 3 countable observable seizures per 4 weeks prior to randomization, including at least the 4-week baseline period.
   2. These seizures may be generalized, focal, or of unknown onset, but may not include absence seizures or focal aware seizures without a detectable motor component, aphasia, or other observable symptom.

      -

Exclusion Criteria:

1. Pregnant or lactating female
2. History of hypersensitivity to ivermectin
3. Ivermectin use within 28 days of screening
4. History of progressive neurological disorder or other significant progressive disorder or unstable medical condition(s)
5. Change in AED regimen in the 28 days prior to screening
6. Taking >4 concomitant AEDs at screening
7. History of status epilepticus in the 2 years prior to screening
8. A vagal nerve stimulator (VNS), responsive neurostimulator (RNS) or deep brain stimulator (DBS), implanted or activated <1 year prior to screening, or with stimulation parameters stable for <3 months or battery life of unit not anticipated to extend for the duration of the trial
9. History of traumatic brain injury within 28 days prior to screening
10. History of psychogenic non-epileptic seizures (PNES), active or within 2 years prior to study entry
11. Epilepsy-related surgery within 1 year prior to screening, epilepsy-related radiosurgery or laser surgery within 1 year prior to screening
12. Epilepsy dietary therapy initiated <3 months prior to screening
13. Psychiatric disorder in which changes in pharmacotherapy are needed or anticipated during the study
14. Active suicidal plan/intent in the 6 months prior to screening and evidenced by a positive response to C-SSRS questions 4 or 5, a history of suicide attempt in the 2 years prior to screening, or more than 1 lifetime suicide attempt.
15. Administration of investigational product in another trial within 28 days prior to the first expected study drug administration, or five half-lives, whichever is longer.
16. Receiving felbamate for <1 year prior to screening
17. Receiving vigabatrin for <2 years prior to screening. Subjects on vigabatrin should have available, appropriate documentation of visual fields
18. Receiving ezogabine (ex-US) at screening
19. Use of the following medications and foods at screening or baseline that may interfere with study drug:

    1. CYP3A4 inducers: rifampin, lumacaftor, mitotane, enzalutamide, apalutamide, St. John's wort, glucocorticoids
    2. CYP3A4 inhibitors including and not limited to: clarithromycin, ceritinib, idelalisib, lonafarnib, tucatinib, erythromycin, telithromycin, diltiazem, ketoconazole, posaconazole, voriconazole, telithromycin, nefazodone, mifepristone, itraconazole, ketoconazole, anti-retroviral drugs (atazanavir, darunavir, indinavir, lopinavir, nelfinavir, ritonavir, saquinavir, tipranavir), grapefruit and grapefruit juice, pomegranate and pomegranate juice
    3. Additional medications that may interact with CYP3A4, PGP, or Vitamin K: fluconazole, isavuconazole, cyclosporine, amiodarone, dronaderone, verapamil, imatinib, warfarin, acenocoumarol
20. Has any of the following laboratory abnormalities at screening:

    1. Positive COVID test
    2. Positive urine drug screen (except as clinically indicated)
    3. Total bilirubin or higher ≥1.5× the site laboratory upper limit of normal (ULN)
    4. ALT or ALT ≥2× the site laboratory ULN
    5. HbA1c >7.0%
    6. Positive hCG (female participants) (screening or baseline)
21. Subject is not approved for study inclusion by the Epilepsy Consortium based on the diagnostic review form
22. Any condition that, in the opinion of the investigator, may impact a subject's safety or ability to follow study procedures.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2022-10-11 (Actual); Study Completion 2023-10-11 (Estimated)

PRIMARY OUTCOMES:
Comparison of Grade 2 or higher, as defined by National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0, November 2017, treatment-related adverse events (TRAEs) in each dose cohort as compared with placebo. | Upto 84 days

SECONDARY OUTCOMES:
Change in C-SSRS responses as compared with baseline in treatment cohort as compared with placebo. | Day 84
Median change in the number of countable seizures overall and by seizure type (focal, generalized, and unknown onset). | Day 14, 42, 70, 98
Median change in the number of generalized tonic-clonic and focal to generalized tonic-clonic seizures. | Day 14, 42, 70, 98
Percent (%) of subjects who are seizure free. | Day 1 upto day 84
Number of subjects who withdraw from treatment because of study-drug effects. | Upto 14 days
Number of subjects in each dose cohort who decrease their dose of study drug because of treatment-related effects. | Upto 14 days
Correlation of plasma levels of EQU-001 with % seizure reduction | Weeks 2, 4, 8, 12
Correlation of plasma levels of biomarkers with % seizure reduction | Weeks 4, 8, 12
Seizure freedom in treated subjects overall and at each dose as compared with placebo. | Weeks 3 to 12 and Weeks 1 to 12 relative to the baseline observation period
Change in the Quality of Life in Epilepsy-31-P (QOLIE-31-P) scale score as compared with baseline in treatment cohort as compared with placebo. | Day 84
  Maximum score: 100, Minimum score: 0, Higher scores reflect better quality of life, lower scores reflect lower quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ya-El Mandel-Portnoy, PhD, Study Director — Equilibre
Locations (10):
- United States (6):
  - Consultants in Epilepsy and Neurology PLLC, Boise, Idaho
  - Mid-Atlantic Epilepsy and Sleep Center, Bethesda, Maryland
  - Northeast Regional Epilepsy Group, Hackensack, New Jersey
  - NYU Langone Medical Center, NYU Comprehensive Epilepsy Center, New York, New York
  - Comprehensive Epilepsy Center at Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Virginia, Charlottesville, Virginia
- Israel (4):
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No